CLINICAL TRIAL: NCT03438604
Title: A Phase 1, 2-Way Crossover Study to Evaluate the Effect of Heat Application on the Delivery Profile of Corplex™ Donepezil 5 mg Transdermal Delivery System (TDS) in Healthy Volunteers
Brief Title: A Study to Evaluate the Effect of Heat Application on the Delivery Profile of Corplex™ Donepezil Transdermal Delivery System (TDS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corium, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P-16039
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Donepezil TDS with Heat Applied (Other): Corplex Donepezil TDS 5 mg/day with heat applied
  Interventions: Drug: Donepezil TDS
- Donepezil TDS without Heat (Other): Corplex Donepezil TDS 5 mg/day with no heat applied
  Interventions: Drug: Donepezil TDS
- Donepezil TDS Extension Study with Heat (Other): Corplex Donepezil TDS 5 mg/day with heat. Two skin sensors will be placed underneath the TDS and adjacent to the TDS.
  Interventions: Drug: Donepezil TDS

INTERVENTIONS:
Drug: Donepezil TDS — Donepezil Hydrochloride Transdermal Delivery System

SUMMARY:
A study to assess the effect of heat application on the delivery profile of Corplex™ Donepezil Transdermal Delivery System (TDS)

DETAILED DESCRIPTION:
2-Way Crossover study

Approximately 24 healthy, adult male and female subjects will be enrolled.

Subjects will be randomized to 1 of 2 treatment sequences prior to the first TDS application in treatment period 1.

For each treatment period, subjects will have one 7-day TDS applied on their back. Depending on which sequence a subject is randomized to, the healthy subject will either be exposed to heat or not during the TDS wear time.

Blood samples for Donepezil PK will be collected pre-dose until the end of each treatment period.

Adhesion will be monitored throughout the TDS wear time, and skin irritation will be monitored after TDS removal.

Subjects who complete the 2-way crossover study may be eligible to participate in the optional Study Extension Period. In the Study Extension Period, subjects will have their skin surface temperature monitored under the patch and adjacent to the TDS.

Blood samples for Donepezil PK will not be collected, and adhesion will not be monitored for the Study Extension TDS wear period.

Safety will be monitored throughout the study by adverse event reporting and repeated clinical and laboratory evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female ≥ 30 years of age

Exclusion Criteria:

* History of any illness that, in the opinion of the investigator, might confound the results of the study or poses an additional risk to the subject by participation in the study
* History or presence of alcoholism or drug abuse within the past 2 years prior to the first study product treatment
* History or presence of hypersensitivity or idiosyncratic reaction to the study products or related compounds
* History of significant multiple and/or severe allergies, or has had an anaphylactic reaction or significant intolerability to prescription or nonprescription drugs
* History or presence of excessive sweating
* History or presence of hairy skin on application sites
* History or presence of significant skin damage or disease at application sites
* Any medical or surgical procedure or trauma within 28 days prior to the first study product treatment

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics, Cmax | Blood samples for donepezil PK will be collected pre-dose until the end of each treatment period, approximately 6 weeks total
  Peak plasma concentration (Cmax) of once-weekly Donepezil TDS in the presence and absence of heat
Pharmacokinetics, AUC | Blood samples for the Donepezil PK will be collected pre-dose until the end of each treatment period, approximately 6 weeks total
  Area under the curve (AUC) of once-weekly Donepezil TDS in the presence and absence of heat

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Daily during 1 week treatment period and during the 5 week follow-on period
  General safety (adverse events and serious adverse events as reported by subject following guidance CTCAE v4.0)
Summary Listing of Skin Irritation Score of Donepezil TDS by post-removal time point | 0.5 hr, 24 hr, 48 hr, 72 hr after each TDS removal (3 days)
  Skin irritation score is determined by the sum of Dermal Response score (8-point categorical scale; where 0=no evidence of irritation to 7=strong reaction) using numeric values and Other Effects score (6-point categorical scale where 0=none observed to H=scabs/erosion) using alphabet letters equivalent to numeric values and summarized by the presence and absence of heat
Application Site Mean Adhesion Scores of Donepezil TDS | Daily during 1 week treatment period
  Adhesion data will be collected during each 7-day patch wear period

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Armas, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
No plans